CLINICAL TRIAL: NCT00541476
Title: Non-Interventional Study In Patients With Peripheral Or Central Neuropathic Pain Undergoing Symptomatic Treatment With Lyrica
Brief Title: Non-Interventional Study In Patients With Peripheral Or Central Neuropathic Pain Treated With Lyrica
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081178
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2008-11

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to obtain more data about efficacy and safety of the study drug Lyrica.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of peripheral or central neuropathic pain

Exclusion Criteria:

* None. Patients recruited by physician decision. Patient's personal data are not collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081178&StudyName=Non-Interventional%20Study%20In%20Patients%20With%20Peripheral%20Or%20Central%20Neuropathic%20Pain%20Treated%20With%20Lyrica